CLINICAL TRIAL: NCT05064176
Title: Comparison of Reconstructive Lymphatic Surgery Versus no Surgery, Additional to Decongestive Lymphatic Therapy (Usual Care), for the Treatment of Iymphoedema, Through a Multicentre Randomised Controlled Trial
Brief Title: Added Value of Reconstructive Lymphatic Surgery to Usual Care in Lymphoedema
Acronym: SurLym
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KCE19-1245
Record Dates: First submitted 2021-08-24; First posted 2021-10-01 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Lymphoedema of Leg; Lymphedema Arm; Lymphedema
Keywords: Reconstructive lymphatic surgery; Decongestive lymphatic therapy; Lymphovenous anastomosis; Lymph node transfer
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Masking Description: Given the nature of the trial, blinding of participants, the person who performs the trial assessments (= investigator) and care providers (surgeon/ physical therapist/ compression specialist) is not feasible.
  The person who will be performing data analyses (= outcome assessor) will be blinded to the participants' randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reconstructive lymphatic surgery (Experimental): The intervention treatment is reconstructive lymphatic surgery and consists of the application of lymphovenous anastomosis (LVA), lymph node transfer (LNT) or a combination of both. The choice of reconstructive technique(s) is determined by the surgeon and is based on the algorithm for reconstructive lymphatic surgery of lymphoedema.
  Additionally, all patients receive usual care (i.e. maintenance decongestive lymphatic therapy)
  Interventions: Other: Usual care; Procedure: Reconstructive lymphatic surgery
- No surgery (Active Comparator): All patients receive usual care (i.e. maintenance decongestive lymphatic therapy)
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Usual care — Home physical therapist performs usual care and educates the patient to perform self-management
  Usual care:
  M1-6: 6 months of maintenance decongestive lymphatic therapy (DLT) (by patient and home physical therapist):
  * week 1-2: no physical therapy; patient performs limb elevation, muscle contractions and wears the bandage (intervention group)/ compression garment (control group)
  * week 3-4: start physical therapy, 2 days/ week: exercises, skin care & manual lymph drainage (MLD), education; self-management by patient and wearing compression garment 14-16h/day (4 sessions) M2-6: 1 day/ week physical therapist: exercises, skin care & MLD, and self-management by patient and wearing compression garment 14-16h/day (20 sessions)
  M7-12: 6 months of maintenance DLT by patient (self-management) and home physical therapist:
  - 1 day/week physical therapist: skin care, MLD, exercises (26 sessions) Month 13-18: 6 months of maintenance DLT by patient Month 19-36: 18 months of follow-up
Procedure: Reconstructive lymphatic surgery — For the procedure of LVA:
  - Aim: making anastomoses of lymph vessels at the capillary level with a diameter of 0.3 to 0.8 mm, to redirect lymph to venous stream directly
  For the procedure of LNT:
  - Aim:
  1. Placed lymph nodes act as sponge to absorb lymphatic fluid and direct it into the vascular network;
  2. Placed lymph nodes induce lymphangiogenesis
  Arms: Reconstructive lymphatic surgery

SUMMARY:
The primary objective of this research proposal is to investigate

* in patients with lymphoedema of the upper limb or lower limb (P)
* the added value of reconstructive lymphatic surgery (I)
* to the decongestive lymphatic therapy (usual care) (C)
* on the lymphoedema-specific quality of life (QoL) (O)
* at 18 months post-surgery/ no surgery (T)

Consequently, a multicentre pragmatic randomised controlled trial is performed to give an answer on following research question: 'Is, in addition to usual care - i.e. decongestive lymphatic therapy -, reconstructive lymphatic surgery (intervention group) superior to no surgery (control group), for the treatment of upper or lower limb lymphoedema?'

DETAILED DESCRIPTION:
Lymphoedema is a chronic and often debilitating condition caused by lymphatic insufficiency. It leads to swelling of the limb and an increased risk of infection. It can be classified as primary (congenital) or secondary (acquired) lymphoedema.

Lymphoedema is very burdensome for the patient and therefore is it often associated with mental problems for example frustration and stress. In addition, because of the increase in volume of the limb, patients also develop physical problems, such as pain, heaviness, loss of strength, and develop functional problems, such as problems with household, mobility or social activities. These mental, physical and functional problems all have a negative impact on quality of life and have an influence on the ability to work. Consensus exist that the first choice of treatment is a conservative treatment. This conservative treatment consists of skin care, compression therapy (i.e. multilayer bandaging and compression garments), exercises and lymph drainage. Reconstructive lymphatic surgery is another option, also often performed: i.e. lymphovenous anastomoses, on the one hand, and a lymph node transfer, on the other hand. By (partially) restoring the lymphatic transport, the reconstructive lymphatic surgery may possibly lead to a larger decrease of the lymphoedema volume and therefore greater discontinuation of the compression garment. Consequently, patients will have an improvement in functioning and quality of life.

Currently, scientific evidence for reconstructive lymphatic surgery for the treatment of lymphoedema is missing. Therefore, the aim of this trial is to investigate the added value of reconstructive lymphatic surgery of the lymphatic system in addition to the conservative treatment, for the treatment of lymphoedema.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral or bilateral, primary or secondary lymphoedema of the upper or lower limb
* If cancer-related lymphoedema, approval for participation in study from oncological specialist (patient participation has to be discussed during Multidisciplinary Oncological Consult); approval if:

  * estimated cancer-related survival is ≥3 years
  * oncological safety is guaranteed: for instance, time interval since radiotherapy/ chemotherapy is ≥3 months
* Lymphoedema stage 1 to 2b
* Objective diagnosis of lymphoedema: ≥ 5% volume difference OR ≥ 2 minor/ 1 major criteria on lymphoscintigraphy OR presence of IndoCyanineGreen (ICG) dermal backflow
* Score on Lymph-ICF questionnaire at screening: ≥ 25 / 100 (= moderate level of problems in functioning related to the development of lymphoedema)
* History of at least 6 months of decongestive lymphatic therapy (DLT) until minimal pitting
* Age ≥ 18 years

Exclusion Criteria:

* Participants with history of liposuction, lymphovenous anastomosis, lymph node transfer
* Pregnant participants
* Severe obese participants: BMI>35
* Estimated cancer-related survival is <3 years and oncological safety is not guaranteed (e.g. interval since radiotherapy/ chemotherapy is <3 months)
* In case of lower limb lymphoedema: presence of chronic venous insufficiency C4, C5, C6; deep venous thrombosis; post-thrombotic syndrome
* Allergy for ICG, iodine, penicillin and sulphonamides; increased activity of thyroid gland; benign tumour in thyroid; heparin use and severe renal insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Lymphoedema-specific QoL (or problems in functioning related to development of lymphoedema) | at 18 months
  evaluated with the Dutch or French version of the Lymph-ICF questionnaire for upper or lower limb lymphoedema

SECONDARY OUTCOMES:
Lymphoedema-specific QoL (or problems in functioning related to development of lymphoedema) | at 1, 3, 6, 12 (short term) and 24, 36 (longer term) months
  evaluated with the Dutch or French version of the Lymph-ICF questionnaire for upper or lower limb lymphoedema
General health-related QoL | at 1, 3, 6, 12, 18, 24, 36 months
  evaluated with the EuroQol-5D-5L questionnaire
Limb volume | at 1, 3, 6, 12, 18 (key secondary outcome), 24, 36 months
  evaluated using circumference measures (ml)
Failure to reduce the hours a day of wearing the compression stocking | at 12, 18, 24, 36 months
  failure is defined as not able to continue the reduction of the hours of wearing the compression garment as stated by the protocol
The hours of wearing the compression garment during one week | at 12, 18 (key secondary outcome), 24, 36 months
  evaluated with the International Compression Club (ICC) questionnaire ('dosage score' between 0-168h)
The experience of the compression garment | at 1, 3, 6, 12, 18, 24, 36 months
  evaluated with the International Compression Club (ICC) questionnaire ('comfort score' between 0-10 and 'complication score' between 0-10)
The physical activity level | at 1, 3, 6, 12, 18, 24, 36 months
  evaluated with the International Physical Activity Questionnaire (IPAQ) - short form (MET-hours/week)
The need for intensive treatment due to an increase in lymphoedema volume | at 6, 12, 18, 24, 36 months
  through interview
Body weight | at 1, 3, 6, 12, 18, 24, 36 months
  measured using a balance
Work capacity | at 1, 3, 6, 12, 18, 24, 36 months
  evaluated with the Work Productivity and Activity Impairment (WPAI-GH) questionnaire
Work ability | at 1, 3, 6, 12, 18, 24, 36 months
  evaluated with the Quickscan 18 (short form) questionnaire
Infection during the previous 18 months (yes/no) | at 18, 36 months (adverse events are collected during each clinical assessment but the amount of infections as secondary outcome are taken together for statistical analyses per 18 months)
  through interview
Complications of surgery | at 1, 3, 6, 12, 18, 24, 36 months
  through interview
Recurrence of cancer (yes/no) | at 36 months
  through medical file
Lymphatic transport | at 18 months
  through lymphoscintigraphy
Costs related to lymphoedema and its treatment during previous 18 months | at 18, 36 months
  through interview

CONTACTS AND LOCATIONS:
Overall Officials: Nele Devoogdt, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Thierry Deltombe, Principal Investigator — CHU-UCL Mont-Godinne; Caren Randon, Principal Investigator — University Hospital, Ghent
Locations (3):
- Belgium (3):
  - Ghent University Hospital, Ghent
  - University Hospitals of Leuven, center for lymphedema, Leuven
  - CHU-UCL Mont-Godinne, Namur

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data (IPD) can be shared upon request.

REFERENCES:
- [Derived] Devoogdt N, De Vrieze T, Heroes AK, Bechter-Hugl B, Fieuws S, Godderis L, Segers K, Maleux G, Deltombe T, Frippiat J, Servaes M, Berners A, Fosseprez P, Krug B, Kayser F, Falticeanu A, Randon C, Monten C, Van Landuyt K, De Pypere B, Degraeve L, Decorte T, De Schryver M, Van Besien V, Devos D, Suominen S, Ayala JM, Pons G, Fourneau I, Thomis S. SurLym trial: study protocol for a multicentre pragmatic randomised controlled trial on the added value of reconstructive lymphatic surgery to decongestive lymphatic therapy for the treatment of lymphoedema. BMJ Open. 2024 May 10;14(5):e078114. doi: 10.1136/bmjopen-2023-078114. PMID 38729754
- See also: Belgium Health Care Knowledge Centre (KCE) — https://kce.fgov.be/en/kce-191245-comparison-of-reconstructive-surgery-versus-no-surgery-additional-to-decongestive
- See also: Improving Care for Edema and Oncology patients (CarEdOn) — https://www.caredon.org/